CLINICAL TRIAL: NCT02826187
Title: Multicentric, Open Label With Retrospective Inclusion and 5 Years Prospective Follow-up of Acetabular Prothetic Implant "Polymax"
Brief Title: Multicentric, Open Label With Retrospective Inclusion and Follow-up of Acetabular Prothetic Implant "Polymax"
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7859
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis
Keywords: Acetabular implant
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acetabular implant: Data to be collected are :
  * Early complications data related to implant or procedure of implantation
  * Late stage complications data
  * Efficacity of treatment with HIP score
  * Patient satisfaction
  * Radiographic evaluation during standard follow-up
  Interventions: Other: Early complications data; Other: Late stage complications data; Other: Patient Satisfaction; Other: Efficacity; Other: Radiographic evaluation

INTERVENTIONS:
Other: Early complications data — Early complications of interest are :
  * New arthroplasty for any reason
  * Related to the implant :
    * Wrong position of the implant
    * Early displacement of the implant
  * Related to the intervention :
    * Hematoma
    * Dislocation (or not causing the resumption of joint replacement)
    * Deep vein thrombosis
    * Pulmonary embolism
    * Acute Infection
Other: Late stage complications data — Late complications taken into account are:
  * New arthroplasty for any reason
  * Aseptic loosening
  * Delayed hypersensitivity reaction type IV
  * Solid Tumors
  * Recurrent dislocation (causing or not the resumption of joint replacement)
  * Allergic reactions of any kind
  * Chronic infection
Other: Patient Satisfaction — Patient satisfaction evaluated by Womac reduced Score
Other: Efficacity — Efficacity as evaluated by Harris HIP score
Other: Radiographic evaluation — Bone reaction visible in radiography

SUMMARY:
Total replacement of hip joint is one of the most important medical innovations of the twentieth century. More than 100,000 hip replacements are being laid each year in France.

Improved fixation, reduced wear rates and reduced implant dislocation rates remain subjects of continuous improvement.

Hip implants cemented and cementless are part of therapeutic arsenal of orthopedic surgeons for joint replacement of the defective hip.

The anchor and friction torque are both essential to the survival of hip implants. Therefore acetabular implants without cement with ceramic insert or polyethylene in a metalback or full polyethylene coated with titanium grains without metalback are proposed, but they have their own complications (Squeaking, fractures, recovery difficulties, difficult radiographic analysis, high cost for ceramics, primary stability defects, instability of the instrument set, Titanium residues in absence of metalback. An alternative to these implants may be an acetabular component without cement with polyethylene insert with an end metalback to increase both polyethylene thickness and size of the head in order to expect a low complication rate with important longevity for a lower cost.

This study was conducted to ensure the safety and effectiveness of the acetabular implant "POLYMAX"

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from hip disease: primary or secondary hip osteoarthritis or osteonecrosis.
* Patient having been implanted with a POLYMAX implant;
* Patient having agreed to participate in a follow-up 5 years;
* Patient who have accepted the use of their data in the context of this study.
* Patient having pre-operative and post-operative data

Exclusion Criteria:

* Pre or post-operative Partial data
* Patients not available for follow up at 2 and 5 years ..
* Metabolic disease or autoimmune witch may interfere with bone growth not allowing the indication of a prosthesis without cement,
* Mental disorder or disease of proven behavior.
* Severe osteoporosis,
* Direct or indirect bone irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Innocuity of POLYMAX acetabular implant as assessed by data collected on early complications | 60 months
Innocuity of POLYMAX acetabular implant as assessed by data collected on late-stage complications | 60 months

SECONDARY OUTCOMES:
Efficacity of POLYMAX acetabular implant as assessed by Harris clinical score | 60 months
Patient satisfaction as assessed by Womac reduced score | 60 months
Evaluation of implant good holding as assessed by apparition of radiolucent lines in radiography | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHIRON, MD, Principal Investigator — University Hospital of Toulouse
Locations (2):
- France (2):
  - Saint Grégoire Hospital, Saint-Grégoire
  - Purpan Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided